CLINICAL TRIAL: NCT06554431
Title: Assessing the Efficacy of Self-Driven Repetitive Artmaking Practice on Pain and Mood States for Patients With Chronic Pain, Opioid Use Disorder, and Opioid Misuse
Brief Title: Assessing the Efficacy of Self-Driven Repetitive Artmaking Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-15440; 1RM1DA055437-01 (NIH)
Record Dates: First submitted 2024-07-25; First posted 2024-08-15 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Opioid Use Disorder; Opioid Misuse; Opioid-Related Disorders
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Repetitive Artmaking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Art Making (Experimental): Each patient will receive artmaking kits
  Interventions: Behavioral: Self-Driven Repetitive Artmaking

INTERVENTIONS:
Behavioral: Self-Driven Repetitive Artmaking — Three (3) art kits which all use repetitive artmaking processes (e.g., materials for mandalas, stamp making kit, weaving kit)

SUMMARY:
The primary purpose of this study is to assess the acceptability of self-directed art making for people with chronic pain and OUD/opioid misuse, or to state it another way, whether people with chronic pain and OUD/opioid misuse will realistically do this artistic practice on their own.

A secondary question of this study is to explore whether doing this art practice can help minimize pain during the artistic process, lessen depression and anxiety, and improve feelings of social connection.

DETAILED DESCRIPTION:
The pilot is an exploratory evaluation of whether repetitive artmaking in home environments is acceptable for chronic pain self-management in individuals with OUD/opioid misuse, and whether self-driven repetitive artmaking can offer respite from pain, depression, and anxiety, and improve social connectivity.

The study will recruit 40 individuals living with chronic pain with an OUD diagnosis or opioid misuse from a Montefiore-led methadone clinic. The Principal Investigators (PIs) will collaborate with an Art Therapist to develop three (3) simple art kits. Patients will participate in an in-person art workshop, to be held in English with the support of a Spanish translator, and complete pre- and post-surveys assessing in-the moment pain, anxiety, depression, and social connectivity. Patients will be given all three (3) kits to take home and to complete the same pre- and post-surveys and art kits at home up to four (4) times within a four-month period to assess real-world adoptability and efficacy. The art kits will not include any visible information about Montefiore or the study in the front of the packets; paper versions of the survey will be enclosed within the kits, to support confidentiality. A subset of patients will be invited to a virtual meaning making group to capture qualitative feedback. The study staff will not share the names of patients with anyone outside the core research team - the co-PIs, Study Coordinator, Patient Advocate, Biostatistician, Art Therapist, and Photographer and Exhibit Coordinator. All patients will be invited to have their art photographed and share their experience of the artmaking process and how it relates to their chronic pain and opioid use.

Photographs and stories will be shared on the Montefiore campus as an art exhibit, and the layperson audience will be surveyed to assess any resultant alteration in feelings of stigma toward the population of those living with chronic pain and OUD/opioid misuse. Patients who share their artwork will be able to decide if their name (or a portion of their name) or a pseudonym will be included in the exhibit alongside their artwork, or whether maintaining anonymity is preferred.

Implementation:

In-Person Workshop: An Art Therapist, will lead three (3) two-hour in-person workshops, with all patients required to attend one (1) in-person workshop as part of this study. Spanish translation will be available at all workshops. The purpose of these workshops are twofold: gather patient characteristic data (demographics, Pain Catastrophizing Survey, questions on experience with art and openness to mindfulness) and orient patients to the use of the art kits available to them to take and use at home. The art therapist will develop three (3) repetitive artmaking kit options and will develop enough for patients to leave the workshop with one of each kit. Options include mandala painting, weaving, and stamp making kits. As previously stated, the art kits will be compiled to minimize visual identification from others that are part of a research study, with all survey materials asking sensitive questions buried in the middle of the packet. At the start of the in-person workshop, PI will orient patients to the pilot goals and activities, answer all questions, collect consent forms, and provide the link to the pre-survey assessing pain and mood as well as paper versions of the survey. The art therapist will provide an engaging overview of the three available kits, and patients will select a kit to try for the in-person workshop. PI will be present to provide Spanish translation and explanation as necessary. The last 15 minutes of the workshop will be saved for patients to complete the post-survey on pain and mood. Finally, patients will be informed that they will be invited to bring their artistic outputs to be photographed by a professional photographer at the end of the four month period and to share their experiences of making the art, so that they can share what they have made with the broader community.

It will be made it clear that displaying their art and sharing their experiences is not mandatory, that patients do not need to decide during the workshop if they will want to share their artwork, and that they will be able to use full, part, or none of their name in the event.

At-Home Artmaking: Patients will be invited to take home all three (3) art kits at the end of the in-person workshop, each of which will allow them to make multiple versions of the type of art in question (i.e., materials for multiple mandalas). Each kit will include printed copies of the pre and post-survey assessing pain and mood, along with a reminder to complete the pre- and post-survey when doing the kits (the end date will be included in the art kits).

Communication from the Survey Coordinator will also include the links to the pre- and post surveys. The instructions will prompt patients to complete the survey immediately before starting the art kit and immediately after concluding. Patients will further be prompted to include a photo of their art in the post-survey and can text their photo to the Study Coordinator if they have phone-based photography capacity. All instructions will be in English and Spanish. This implementation process is designed to assess real-world use of the art kits.

The pilot study is an exploratory implementation and mixed methods evaluation of self-guided repetitive art-making to assess the impact of this artistic practice on:

1. self-reported pain levels,
2. self-reported mood states including anxiety and depression, and
3. self-reported feelings of connection for patients living with chronic pain and opioid use disorder (OUD) or documented misuse of opioids.

A secondary research focus will be to assess whether viewing art made by patients with chronic pain and OUD/opioid misuse diminishes stigma towards these populations for the broader population.

Aim 1 (Acceptability): Develop three (3) self-guided repetitive artmaking kits for patients with chronic pain and OUD/opioid misuse to use on their own, with instructions in English and Spanish, and train the patients on the use of these artmaking kits through three (3) in person workshops in English and Spanish.

Hypothesis 1: Simple art kits that offer repetitive artmaking practices will be acceptable for and interesting to patients with chronic pain and OUD/opioid misuse. Acceptability will be measured as described in the Outcome Measures. Brief questions will be asked at the workshops to assess patients' previous experience with art and openness to mindfulness activities, along with a brief demographic questionnaire, to provide a baseline.

Aim 2 (Efficacy): Evaluate whether the self-guided repetitive artmaking kits significantly impact patients' self-reported experiences of pain, mood (inclusive of depression and anxiety), and social isolation.

Hypothesis 2: Repetitive artmaking will reduce experiences of pain for patients with both chronic pain and OUD/opioid misuse. Significant pain reduction during artmaking practice as captured using the first three questions of the Brief Pain Inventory (BPI) Reduced Minus Peg Questions 8-item questionnaire - questions one and two will be only asked in the pre-survey as these questions ask about pain over the last week and will therefore not change before and after a solo artmaking experience. Patients will also complete the 6-item Pain Catastrophizing Questionnaire as described in the Outcome Measures. This data will be supplemented with qualitative data from the meaning making session and storytelling content, for those who participate.

Hypothesis 3: Repetitive artmaking will reduce depression and anxiety and improve mood for patients with chronic pain and OUD/opioid misuse as described in the Outcome Measures. This data will be supplemented with qualitative data from the meaning making session and storytelling content, for those who participate.

Hypothesis 4: Supporting patients with chronic pain and OUD/opioid misuse in making art will result in higher ratings of social connectivity. Significant improvement in social connectivity during artmaking practice will be captured using the IOS-CC and assessed as described in the Outcome Measures.

Hypothesis 5: Repetitive artmaking will reduce opioid misuse in patients. Any reduction in non-prescribed opioid use as captured as described in the Outcome Measures. This data will be supplemented with qualitative data from the meaning making session and storytelling content, for those who participate.

Aim 3 (Community Intervention): Prepare an exhibit of art made by patients and stories of their experiences and evaluate whether this exhibit impacts stigma regarding chronic pain and opioid use in the broader population (audience).

Hypothesis 6: Laypersons viewing photographs of the art paired with patients' descriptions of their art and the artmaking process, will lessen stigma towards people with chronic pain and OUD/opioid misuse. Laypersons who view the exhibit and who complete a retroactive pre-post survey will self-report lessened stigma towards persons with chronic pain and OUD/opioid misuse through positive appraisal of the artists. This data will be supplemented with qualitative data from the meaning making session and storytelling content, for those who participate.

ELIGIBILITY:
Inclusion Criteria:

1. Experience chronic pain
2. Have received medication for OUD in the past 30 days or meet criteria for opioid misuse
3. Are aged 18 or older
4. Are fluent in English and/or Spanish

Exclusion Criteria:

1. Are not fluent in either English or Spanish
2. Are unable to participate in and complete the introductory workshop due to language or other barriers - physical disabilities are not exclusionary
3. Do not otherwise meet the inclusion criteria for age, OUD, Opioid misuse, and chronic pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Intervention | 4 months
  Feasibility of the intervention will be measured quantitatively by the number of patients who complete the pre- and post-survey up to four (4) times. Group mean results will be summarized.
Acceptability of the Intervention | 4 months
  Acceptability of the intervention will be measured during listening sessions with participants responding to questions regarding whether they used the art kits at home AND whether they report to the Study Coordinator (SC) during monthly check-ins to confirm that they have engaged with the art kits on their own. Group mean results will be summarized using basic descriptive statistics.

SECONDARY OUTCOMES:
Mood outcomes - Anxiety | Before and after a microintervention within a 24 hour period, up to 4 months
  Anxiety before and after the workshop and each instance of repetitive art making (up to 4 sessions) will be assessed based on a single question administered during the survey: "How anxious are you feeling right now?" Patient responses will be scored on a 5-point Likert scale ranging from 0 ("Extremely") to 4 ("Not at all"). In this context, higher scores are associated with reduced levels of worrying and fearfulness regarding everyday situations. Group results will be summarized using basic descriptive statistics.
Mood outcomes - Depression | Before and after a microintervention within a 24 hour period, up to 4 months
  Depression before and after the workshop and each instance of repetitive art making (up to 4 sessions)will be assessed based on a single question administered during the survey: "How sad are you feeling right now?" Patient responses will be scored on a 5-point Likert scale ranging from 0 ("Extremely") to 4 ("Not at all"). In this context, higher scores are associated with reduced levels of feeling down or hopelessness and increased pleasure in daily activities. Group results will be summarized using basic descriptive statistics.
Current Level of Pain | Before and after a microintervention within a 24 hour period, up to 4 months
  Current level of pain before and after the workshop and each instance of repetitive art making (up to 4 sessions) will be assessed based on a single question administered during the survey. Patients will be asked to rate the severity of their current pain on a scale ranging from 0 ("No Pain") to 10 = ("Pain as bad as you can imagine") with higher scores being associated increased pain severity. Group results will be summarized using basic descriptive statistics.
Previous week pain - at its worst | Before the workshop and before each microintervention within a 24 hour period, up to 4 months
  Previous week pain (at its worst) will be assessed before the workshop and before each instance of repetitive art making (up to 4 sessions) by asking patients a single question to describe the least and most pain they have experienced over past week (7 days) on a scale ranging from 0 ("No Pain") to 10 ("Pain as bad as you can imagine") with higher scores being associated increased pain severity. Group results will be summarized using basic descriptive statistics.
Previous week pain - at its least | Before the workshop and before each microintervention within a 24 hour period, up to 4 months
  Previous week pain (at its least) will be assessed before the workshop and before each instance of repetitive art making (up to 4 sessions) by asking patients a single question to describe the least and most pain they have experienced over past week (7 days) on a scale ranging from 0 ("No Pain") to 10 ("Pain as bad as you can imagine") with higher scores being associated increased pain severity. Group results will be summarized using basic descriptive statistics.
Pain Experiences | Before the workshop, within 24 hours
  Pain experiences before the workshop will be assessed based on patient responses on the 6-item Pain Catastrophizing Scale (PCS-6) conducted during the in-person workshop. The PCS-6, a short form of the PCS questionnaire, consists of six statements (Items 4, 5, 6, 10, 11, and 13 from the 13-item PCS questionnaire) which ask about the degree of pain catastrophizing on a 5-point Likert scale ranging from 0 ("Not at all") to 4 ("All the time") for an overall possible scoring range of 0-24. Higher scores are associated with increased perceptions of helplessness regarding their pain, magnification of their pain, and pain-related rumination. Group results will be summarized using basic descriptive statistics.
Social Connectivity | Before and after a microintervention within a 24 hour period, up to 4 months
  Social Connectivity before and after the workshop and each instance of repetitive art making (up to 4 sessions) will be assessed using the Inclusion of Other in the Self Scale to assess Communal Coping (IOS-CC). Patients are presented with seven pairs of circles that range from just touching to almost completely overlapping. One circle in each pair is labeled "self," and the second circle is labeled "other." Patients are asked to choose the pair of circles that best describe their relationship to their community. Responses are scored as: 1 = no overlap; 2 = little overlap; 3 = some overlap; 4 = equal overlap; 5 = strong overlap; 6 = very strong overlap; 7 = most overlap such that the higher the score the stronger the bond with their community. Group results will be summarized using basic descriptive statistics.
Non-prescribed Opioid Use | Before and after a microintervention within a 24 hour period, up to 4 months
  Non-prescribed opioid use before and after the workshop and each instance of repetitive art making (up to 4 sessions) will be assessed based on a response to a binary question (modified from the Addiction Severity Index) as to whether the patient has used non-prescription opioids during the past 24 hours. "No" responses will be assigned a score of 0; "Yes" responses will be assigned a score of 1. Group results will be summarized.
Level of Opioid Highness | Before and after a microintervention within a 24 hour period, up to 4 months
  Level of opioid highness before and after the workshop and each instance of repetitive art making (up to 4 sessions) will be assessed based on a single question derived from the modified, Daily Sessions, Frequency, Age of Onset, and Quantity of Cannabis Use (DFAQ-CU) inventory with the exception that the question is focused on opioids not cannabis. Patients will be asked to share how high they are at the time of the survey on a 5-point Likert scale ranging from 0 ("I am not high") to 4 ("I am very high") such that higher scores are associated with increased states of being high. Group results will be summarized using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Seham, PhD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Wellness Center at Waters Place, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yong RJ, Mullins PM, Bhattacharyya N. Prevalence of chronic pain among adults in the United States. Pain. 2022 Feb 1;163(2):e328-e332. doi: 10.1097/j.pain.0000000000002291. PMID 33990113
- [Background] Rikard SM, Strahan AE, Schmit KM, Guy GP Jr. Chronic Pain Among Adults - United States, 2019-2021. MMWR Morb Mortal Wkly Rep. 2023 Apr 14;72(15):379-385. doi: 10.15585/mmwr.mm7215a1. PMID 37053114
- [Background] Lerman SF, Rudich Z, Brill S, Shalev H, Shahar G. Longitudinal associations between depression, anxiety, pain, and pain-related disability in chronic pain patients. Psychosom Med. 2015 Apr;77(3):333-41. doi: 10.1097/PSY.0000000000000158. PMID 25849129
- [Background] Fishbain DA, Cutler R, Rosomoff HL, Rosomoff RS. Chronic pain-associated depression: antecedent or consequence of chronic pain? A review. Clin J Pain. 1997 Jun;13(2):116-37. doi: 10.1097/00002508-199706000-00006. PMID 9186019
- [Background] Allen SF, Gilbody S, Atkin K, van der Feltz-Cornelis C. The associations between loneliness, social exclusion and pain in the general population: A N=502,528 cross-sectional UK Biobank study. J Psychiatr Res. 2020 Nov;130:68-74. doi: 10.1016/j.jpsychires.2020.06.028. Epub 2020 Aug 1. PMID 32791383
- [Background] McCaffrey R, Frock TL, Garguilo H. Understanding chronic pain and the mind-body connection. Holist Nurs Pract. 2003 Nov-Dec;17(6):281-7; quiz 288-9. doi: 10.1097/00004650-200311000-00002. PMID 14650569
- [Background] Angheluta A-M., & Lee, B. L. (2011). Art therapy for chronic pain: Applications and future directions. Canadian Journal of Counselling and Psychotherapy, 45(2), 112-131.
- [Background] Dahlhamer JM, Connor EM, Bose J, Lucas JL, Zelaya CE. Prescription Opioid Use Among Adults With Chronic Pain: United States, 2019. Natl Health Stat Report. 2021 Aug;(162):1-9. PMID 34524076
- [Background] Keyes KM, Rutherford C, Hamilton A, Barocas JA, Gelberg KH, Mueller PP, Feaster DJ, El-Bassel N, Cerda M. What is the prevalence of and trend in opioid use disorder in the United States from 2010 to 2019? Using multiplier approaches to estimate prevalence for an unknown population size. Drug Alcohol Depend Rep. 2022 Jun;3:100052. doi: 10.1016/j.dadr.2022.100052. Epub 2022 Apr 8. PMID 35783994
- [Background] Substance Abuse and Mental Health Services Administration (SAMHSA). (2021). Highlights for the 2021 National Survey on Drug Use and Health. Retrieved May 22, 2023 from https://www.samhsa.gov/datasites/default/files/2022- 12/2021NSDUHFFRHighlights092722.pdf
- [Background] Premier, Inc. (2019, January 30). Opioid overdoses costing U.S. hospitals an estimated $11 billion annually. Retrieved May 22, 2023 from https://www.premierinc.com/newsroom/press-reoleases/opioid-overdoses/costing-u-shospitals-an-estimated-11-billion-annually
- [Background] Florence C, Luo F, Rice K. The economic burden of opioid use disorder and fatal opioid overdose in the United States, 2017. Drug Alcohol Depend. 2021 Jan 1;218:108350. doi: 10.1016/j.drugalcdep.2020.108350. Epub 2020 Oct 27. PMID 33121867
- [Background] Shella, T. A. (2018). Art therapy improves mood, and reduces pain and anxiety when offered at bedside during acute hospital treatment. The Arts in Psychotherapy, 57, 59-64.
- [Background] Hass-Cohen N., Bokoch, R., Goodman, K., & Conover, K. J. (2021). Art therapy drawing protocols for chronic pain: Quantitative results from a mixed method pilot study. The Arts in Psychotherapy, 73, 101479.
- [Background] Angheluta A-M., & Lee, B. L. (2011). Art therapy for chronic pain: Applications and future directions. Canadian Journal of Counselling and Psychotherapy, 45(2), 112-131
- [Background] American Art Therapy Association. (2008). About art therapy. Retrieved May 22, 2023 from https://arttherapy.org/about-art-therapy/
- [Background] Bullington, J., Nordemar, K., Nordemar, R., & Sjöström-Flanagan, C. (2005). From pain through chaos to new meaning: Two case studies. The Arts in Psychotherapy, 32, 261-274.
- [Background] Pavlek, M. (2008). Paining out: An integrative pain therapy model. Clinical Social Work Journal, 36 385-393.
- [Background] Sivik T, Schoenfeld R. Psychosomatic integrative treatment and rehabilitation. Adv Mind Body Med. 2005 Fall-Winter;21(3-4):55-8. No abstract available. PMID 20671349
- [Background] Long, J. L. (2004). Medical art therapy: Using imagery and visual expression in healing. In P. Camic & S. Knight (Eds.). Clinical handbook of health psychology: A practical guide to effective interventions (2nd ed., pp. 315-341). Toronto ON: Hogrefe & Huber.
- [Background] Shapiro B. (1985). All I have is pain: Art therapy in an inpatient chronic pain relief unit. American Journal of Art Therapy, 24(2), 44-48.
- [Background] Burns P, Van Der Meer R. Happy Hookers: findings from an international study exploring the effects of crochet on wellbeing. Perspect Public Health. 2021 May;141(3):149-157. doi: 10.1177/1757913920911961. Epub 2020 Apr 3. PMID 32245337
- [Background] Collen M. Life of pain, life of pleasure: pain from the patients' perspective--the evolution of the PAIN exhibit. J Pain Palliat Care Pharmacother. 2005;19(4):45-52. PMID 16431832
- [Background] Reynolds F, Prior S. 'A lifestyle coat-hanger': a phenomenological study of the meanings of artwork for women coping with chronic illness and disability. Disabil Rehabil. 2003 Jul 22;25(14):785-94. doi: 10.1080/0963828031000093486. PMID 12959359
- [Background] Langarten H. B. (19871). Clinical art therapy: A comprehensive guide. New York, NY: Brunner/Mazel.
- [Background] Dannecker, K. (1991). Body and expression: Art therapy with rheumatoid patients. American Journal of Art Therapy, 29(4), 110-118.
- [Background] Feen-Calligan, H., Washington, O. G. M., & Moxley, D. P. (2008). Use of artwork as a visual processing modality in group treatment of chemically dependent minority women. The Arts in Psychotherapy, 35, 287-295.
- [Background] Holt, E., & Kaiser, D. H. (2009). The first step series: Art therapy for early substance abuse treatment. The Arts in Psychotherapy, 36, 245-250.
- [Background] Schmanke, L. (2017). Art therapy and substance abuse: Enabling recovery from alcohol and other drug addiction. London, UK: Jessica Kingsley Publishers.
- [Background] Skeffington, P. M., & Browne, M. (2014). Art therapy, trauma and substance misuse: Using imagery to explore difficult past with a complex client. International Journal of Art Therapy, 19(3), 114-121.
- [Background] Leis JA, Morrison CI. An Integrative Review of Arts-Based Strategies for Addressing Pain and Substance Use Disorder During the Opioid Crisis. Health Promot Pract. 2021 May;22(1_suppl):44S-52S. doi: 10.1177/1524839921996065. PMID 33942641
- [Background] Stasny, A. (2022). The opioid epidemic and the need for arts in community based treatment options: A literature review. [Thesis, Lesley University].
- [Background] Butler, D. & Moseley, L. (2008). Explain pain. Adelaide, Australia: NOI Group.
- [Background] Cudill, M. A. (2002). Managing pain before it manages you. New York, NY: Guilford.
- [Background] Stinley, N. E., Norris, N. O., & Hinds, P. S. (2015). Creating mandalas for the management of acute pain symptoms in pediatric patients. Art Therapy, 32(2), 46-53.